CLINICAL TRIAL: NCT04809831
Title: A Comparison Between Biorepair Peribioma Toothpaste and Mousse Versus Chlorhexidine 0,2% Toothpaste (Curasept Trattamento Rigenerante) for Domiciliary Oral Care in Periodontal Patients.
Brief Title: The Use of Biorepair Peribioma Toothpaste and Mousse for Home Oral Care in Patients Undergoing Periodontal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Research Resident, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-PERIBIOMA
Record Dates: First submitted 2021-03-16; First posted 2021-03-22 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Periodontal Diseases
Keywords: dental hygiene; periodontal non-surgical therapy; split-mouth
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: This is a study in which patients are divided into two groups:
  * Trial Group: professional dental hygiene at T0, T1 and T2 + Biorepair Peribioma Toothpaste and Mousse for domiciliary oral care twice a day until T2;
  * Control Group: professional dental hygiene at T0, T1 and T2 + Curasept Toothpaste with chlorhexidine 0,2% twice a day until T2.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial Group - Biorepair Peribioma Toothpaste + Mousse (Active Comparator): Domiciliary oral hygiene with Biorepair Peribioma Toothpaste in association with Peribioma Mousse twice a day until T2 session.
  Interventions: Other: Domiciliary oral care with Biorepair Peribioma Toothpaste + Mousse
- Control Group - Curasept Toothpaste (chlorhexidine 0,2%) (Active Comparator): Domiciliary oral care with Curasept Toothpaste (chlorhexidine 0,2%) twice a day until T2 session.
  Interventions: Other: Domiciliary oral care with Curasept Toothpaste (chlorhexidine 0,2%)

INTERVENTIONS:
Other: Domiciliary oral care with Biorepair Peribioma Toothpaste + Mousse — Patients will use Biorepair Peribioma Toothpaste and Mousse for domiciliary oral hygiene twice a day until T2 session.
  Arms: Trial Group - Biorepair Peribioma Toothpaste + Mousse
Other: Domiciliary oral care with Curasept Toothpaste (chlorhexidine 0,2%) — Patients will use Curasept Toothpaste (chlorhexidine 0,2%) for domiciliary oral hygiene twice a day until T2 session.
  Arms: Control Group - Curasept Toothpaste (chlorhexidine 0,2%)

SUMMARY:
This is a split-mouth randomized clinical trial in which a new domiciliary oral care protocol with Biorepair Peribioma Toothpaste and Mousse is evaluated in periodontal patients.

DETAILED DESCRIPTION:
This is a split-mouth randomized clinical trial that aims to suggest an innovative protocol for domiciliary oral care of periodontal patients. In details, home use of Biorepair Peribioma Toothpaste and Mousse is proposed as a support of professional hygiene sessions.

Patients that respond to the eligibility criteria and that sign the informed consent are recruited for periodontal therapy.The first professional hygiene session is performed at the baseline (T0); the following ones will be performed after 3 (T1) and 6 months (T2) from the baseline. In each session, periodontal indices of inflammation are detected; then, subgingival removal of plaque and tartar is performed, followed by glycine air-flow application in periodontal pockets. A microbiological test is perfomed in order to detect red and orange complex bacteria. At this time, patients are randomly allocated into two groups:

* Trial Group: domiciliary oral hygiene with Biorepair Peribioma Toothpaste and Mousse twice a day until T2 session.
* Control Group: home oral hygiene with Curasept Toothpaste (0,2% Chlorhexidine) twice a day until T2 session.

At the end of T1 and T2 professional session, a satisfaction survey about Peribioma Toothpaste and Mousse will ben given to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Presence of periodontal disease according to the recent 2017 classification (2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions): severity grade II-III and complexity grade I-II.
* Presence of bilateral periodontal probes, for at least one tooth per side up to 20 elements with pathologic probes).
* Patients' good compliance

Exclusion Criteria:

* Patients with cardiac pacemaker
* Patients suffering from neurological disorders
* Patients suffering from psychological disorders
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Change in BOP - Bleeding on Probing (percentage) | 3 and 6 months.
  Site-specific assessment of the presence or absence of gum bleeding after the insertion of the periodontal probe for the detection of PPD, detected on 6 sites.
  Percentage of sites with bleeding on probing determines the BOP%.
Change in BS - Bleeding Score | 3 and 6 months.
  Scoring criteria:
  * 0 = no bleeding;
  * 1 = punctiform bleeding in the site of probing;
  * 2 = slightly extended bleeding in the site of probing;
  * 3 = bleeding in more than a half of gingival margin;
  * 4 = gingival border fully covered by blood.
Change in SBI - Sulculus Bleeding Index (Muhulemann and Son, 1781) | 3 and 6 months.
  Scoring criteria:
  * 0 = healthy looking papillary and marginal gingiva, no bleeding on probing;
  * 1 = healthy looking gingiva, with bleeding on probing;
  * 2 = bleeding on probing, change in color, no edema;
  * 3 = bleeding on probing, change in color, slight edema;
  * 4 = bleeding on probing, change in color, obvious edema;
  * 5 = spontaneous bleeding, change in color, marked edema.
Change in GI - Gingival Index (Loe and Silness, 1963) | 3 and 6 months.
  Scoring criteria:
  * 0 = normal gingiva.
  * 1 = mild inflammation, edema and swelling; no bleeding.
  * 2 = moderate inflammation with edema, swelling and bleeding on probing.
  * 3 = severe inflammation with marked edema, redness tissues, ulceration and spontaneous bleeding.
Change in PPD - Probing Pocket Depth | 3 and 6 months.
  Evaluation (in mm) of the depth of the gingival sulcus, through a millimeter periodontal probe; it is detected from the gingival margin to the bottom of the gingival sulcus or periodontal pocket, evaluated at 6 sites.
Change in CAL - Clinical Attachment Loss | 3 and 6 months.
  Measurement (in mm) of the position of the gingival margin in relation to the cemento-enamel junction (CEJ).
Change in Percentage of pathological sites | 3 and 6 months.
  Evaluation of the presence of pathological probes expressed as a percentage.
Change in R - Gingival recession | 3 and 6 months.
  Distance (in mm) between the gingival margin and the amelo-cemental junction.
Change in PI - Plaque Index (Silness and Löe, 1964) | 3 and 6 months.
  Scoring criteria:
  * 0 = no plaque;
  * 1 = thin plaque layer at the gingival margin, only detectable by scraping with a probe;
  * 2 = moderate layer of plaque along the gingival margin; interdental spaces free, but plaque is visible to the naked eye;
  * 3 = abundant plaque along the gingival margin; interdental spaces filled with plaque.
Change in Evaluation of the total height of the adherent gingiva | 3 and 6 months.
  Evaluation (in mm) of the total height of adherent gingiva.
Change in API - Approximal Plaque Index (Lange, 1986) | 3 and 6 months.
  Following application of disclosing, a simple yes/no decision is made concerning whether the interproximal surfaces are covered by plaque (+) or not (-). The proportion of plaque-covered interproximal spaces is expressed as a percentage. Usually, in a given quadrant the interproximal spaces are scored from only one aspect (i.e. from the facial - Q2 and Q4 - or from the oral aspect - Q1 and Q3).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD., Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to Principal Investigator.